CLINICAL TRIAL: NCT01120769
Title: Acetaminophen to Prevent Ischemic Oxidative Reperfusion Injury During Percutaneous Coronary Intervention for Acute Myocardial Infarction
Acronym: APRIORI Pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issue
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, John Oates, Professor of Medicine, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 100001
Record Dates: First submitted 2010-05-06; First posted 2010-05-11 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Acute Myocardial Infarction
Keywords: Myocardial Infarction; Percutaneous Coronary Intervention; Acetaminophen; Lipid Peroxidation
MeSH Terms: conditions — Myocardial Infarction | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen (Active Comparator)
  Interventions: Drug: Acetaminophen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen — single dose
  Arms: Acetaminophen
Drug: Placebo — single dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the hypothesis that acetaminophen will reduce lipid peroxidation and isoprostane formation during reperfusion after percutaneous revascularization for acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

- Patients presenting with STEMI

Exclusion Criteria:

* Duration of symptoms > 12 hours
* Suspected LM or proximal LAD occlusion (based on EKG interpretation)
* Hemodynamic instability
* Acetaminophen use in prior 24 hours
* Use of dipyridamole, or Aggrenox, a formulation of aspirin and extended-release dipyridamole, within 48 hours
* Current use of the following medications: phenytoin, valproic acid, phenobarbital, topiramate, rifampin, carbamazepine, cyclophosphamide, ritonavir, efavirenz, St. John's Wort
* Chronic heavy alcohol use
* Chronic liver disease (other than non-alcoholic fatty liver infiltration)
* Severe valvular heart disease
* Stroke in the past 60 days
* Active major bleeding
* Major surgery in the past 30 days
* Ongoing treatment for active malignancy
* Life expectancy less than 12 months as determined by the patient's attending physician
* Pregnancy
* asthma or severe COPD
* active wheezing on presentation
* allergy or prior adverse reaction to adenosine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Plasma isoprostane level | 60 minutes

SECONDARY OUTCOMES:
Index of microcirculatory resistance | Average 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States